CLINICAL TRIAL: NCT00034151
Title: A Phase IIA Evaluation of Safety and Efficacy of Weekly S-8184 Paclitaxel Injectable Emulsion in Second Line Treatment of Stage III or IV Platinum Resistant Ovarian Cancer or Primary Peritoneal Carcinoma
Brief Title: Safety and Efficacy of S-8184 in Second Line Treatment of Stage III or IV Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Monica Krieger, VP Regulatory Affairs, OncoGenex Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SON-8184-1061
Record Dates: First submitted 2002-04-23; First posted 2002-04-24 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

INTERVENTIONS:
Drug: S-8184 Paclitaxel Injectable Emulsion

SUMMARY:
Phase IIA, multicenter, dose escalation study evaluating the safety and efficacy of weekly S-8184 paclitaxel injectable emulsion in second line treatment of patients with stage III or IV platinum resistant ovarian cancer or primary peritoneal carcinoma.

DETAILED DESCRIPTION:
The goals of this study are to determine the objective response rate, to determine time to disease progression, duration of response, and survival, and to identify the maximum tolerated weekly dose and principal toxicities of S-8184 in this patient population.

ELIGIBILITY:
Inclusion Criteria:

Histologic diagnosis of ovarian cancer or primary peritoneal carcinoma

Stage III or IV disease

One and only one prior cytotoxic chemotherapy regimen which must have included a platinum agent

Platinum resistant disease, defined as documented progression within six months of completion of first line therapy

Adult (18 years of age or older) patients

Adequate hematologic function (ANC greater than 1500 cells/mm3 and platelets greater than 100,000/mm3)

Serum creatinine less than 2.0 mg/dL

Total bilirubin less than 1.5 mg/dL; SGOT and SGPT less than 3 times the upper limit of institutional normal values

ECOG performance status of 0 - 2

Bidimensional measurable or clinically evaluable disease

Patients who have signed an IRB / Ethics Committee approved informed consent

Life expectancy at least 12 weeks

Patient has fully recovered from any previous surgery (at least 4 weeks since major surgery)

Patient has a negative pregnancy test prior to study entry if premenopausal. (Patients of child bearing potential must use a medically effective form of contraception during the treatment.)

Exclusion Criteria:

Patients who have received any taxane-containing preparation including Taxol (paclitaxel) or Taxotere (docetaxel)

Females who are pregnant or lactating

Patients with peripheral neuropathy NCI-CTC grade 2 or greater

Patients who have received wide-field radiation, cytotoxic chemotherapy or hormonal therapy within 4 weeks of study entry; or mitomycin or nitrosoureas within 6 weeks of study entry

Patients who have had an investigational agent within 4 weeks of study entry

Patients receiving concurrent anticonvulsants known to induce P450 isoenzymes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2002-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Determine the objective and partial response rates | No time frame-based on number of patients

SECONDARY OUTCOMES:
Time to progression, duration of response and duration of survival | Based on number of patients